CLINICAL TRIAL: NCT00006310
Title: KSHV Seroprevalence in Hospital Patients From San Antonio
Brief Title: KSHV Infection in Blood Donors From Texas
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 918; R01HL060604 (NIH)
Record Dates: First submitted 2000-09-28; First posted 2000-09-29 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Blood Donors; Acquired Immunodeficiency Syndrome; Blood Transfusion; Herpesvirus, Kaposi Sarcoma-Associated; Sarcoma, Kaposi; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sarcoma, Kaposi; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine the seroprevalence of Kaposi's sarcoma-associated herpesvirus (KSHV/HHV8) in blood donors from Texas. Also to examine the donors' demographic characteristics and to characterize the KSHV using polymerase chain reaction.

DETAILED DESCRIPTION:
BACKGROUND:

Kaposi's sarcoma-associated herpesvirus (KSHV/HHV8) is a blood-borne virus that is etiologically associated with Kaposi's sarcoma (KS), primary effusion lymphoma which is a form of non-Hodgkin's lymphoma, and a subset of multicentric Castleman's disease which is a lymphoproliferative disorder. The investigators developed serologic assays to measure antibodies specific to KSHV latent and lytic antigens. Antibodies to KSHV antigens are found in 70-100 percent of all clinical forms of KS patients. In contrast, relatively low prevalence (2 to 5 percent) is found in the general population of North America. Seroconversion is detected prior to KS onset in AIDS-KS patients, suggesting that primary KSHV infection occurs predominantly in adulthood and is not ubiquitous. Antibody titers to KSHV antigens remain elevated for years after seroconversion. The investigators have recently found a 5 percent prevalence of KSHV infection in blood donors from San Antonio. Further, KSHV has been found in the peripheral blood mononuclear cells (PBMC) of blood donors, and organ transplantation and animal studies have provided evidence of likely person-to-person transmission of KSHV. Thus, KSHV is a potential candidate for screening in blood and plasma donors in view of its etiologic role for several malignancies, low but appreciable prevalence in the general population, and lifelong persistence in a cross-sectional study in blood donors from Texas.

DESIGN NARRATIVE:

The first aim of the study was to determine the prevalence of KSHV infection in blood donors using specific KSHV serologic assays. The investigators used recently developed KSHV specific serologic assays for detecting antibody to KSHV latent nuclear antigen, lytic antigen, and orf65 (lytic antigen minor capsid protein) to determine the prevalence of KSHV infection in a cross-sectional study of four representative blood banks in San Antonio, Dallas, and Houston, Texas. A total of 500 random donors at each site were studied to detect site-specific seroprevalence to plus or minus 2 percent with 95 percent confidence.

The second aim of the study was to analyze the demographic characteristics and the patterns of other blood-borne infections of KSHV-seropositive blood donors. The cross-sectional study in Houston and San Antonio was expanded to prospective study seroprevalence in a larger population with questionnaire obtained demographic data to include gender, age, ethnicity, education level, household income, and zip code. A total of 10,500 donors were obtained from Houston. As the San Antonio center had the highest proportion of Hispanic donors, an additional 2,000 donors were obtained and characterized demographically.

The third aim was to investigate KSHV molecular epidemiology in blood donors through sequence determination of specific nested-polymerase chain reaction (PCR) and RT-PCR products from peripheral blood mononuclear cells (PBMC) of KSHV-seropositive donors. The 2,000 blood samples from San Antonio were also used to amplify KSHV sequences from peripheral blood mononuclear cells of KSHV positive donors using PCR, nested PCR and RT-PCR with and without phorbol ester induction. Sequencing of amplified products was compared to KSHV isolates from New York, Italy, England, and Africa for phylogenetic analysis and assessment of diversity and distribution of KSHV strains in Texas. While the proposed sampling represented only one center in Texas, comparison to isolates for New York and abroad allowed determination of the likelihood that Texas strains were unique or imported from Europe or Africa.

This regional project was performed in collaboration with the University Health System Donor Center in San Antonio, BloodCare in Dallas, and Gulf Coast Regional Blood Center in Houston, thus providing results for three separate metropolitan areas with rather different ethnic compositions. These studies should provide valuable information to assess the necessity and feasibility of national screening of blood donors for KSHV, and gain insight into the patterns of infection as well as the diversity, the distribution, and the origins of the virus strains in blood donors.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-04; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: Shou-Jiang Gao, PhD, Principal Investigator — University of Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang XP, Zhang YJ, Deng JH, Pan HY, Zhou FC, Montalvo EA, Gao SJ. Characterization of the promoter region of the viral interferon regulatory factor encoded by Kaposi's sarcoma-associated herpesvirus. Oncogene. 2001 Jan 25;20(4):523-30. doi: 10.1038/sj.onc.1204115. PMID 11313983
- [Background] Zhang YJ, Deng JH, Rabkin C, Gao SJ. Hot-spot variations of Kaposi's sarcoma-associated herpesvirus latent nuclear antigen and application in genotyping by PCR-RFLP. J Gen Virol. 2000 Aug;81(Pt 8):2049-2058. doi: 10.1099/0022-1317-81-8-2049. PMID 10900044
- [Background] Oyajobi BO, Deng JH, Dallas SL, Jenson HB, Mundy GR, Gao SJ. Absence of herpesvirus DNA sequences in the 5T murine model of human multiple myeloma. Br J Haematol. 2000 May;109(2):413-9. doi: 10.1046/j.1365-2141.2000.02038.x. PMID 10848833
- [Background] Zhang YJ, Davis TL, Wang XP, Deng JH, Baillargeon J, Yeh IT, Jenson HB, Gao SJ. Distinct distribution of rare US genotypes of Kaposi's sarcoma-associated herpesvirus (KSHV) in South Texas: implications for KSHV epidemiology. J Infect Dis. 2001 Jan 1;183(1):125-9. doi: 10.1086/317650. Epub 2000 Nov 30. PMID 11106539
- [Background] Baillargeon J, Deng JH, Hettler E, Harrison C, Grady JJ, Korte LG, Alexander J, Montalvo E, Jenson HB, Gao SJ. Seroprevalence of Kaposi's sarcoma-associated herpesvirus infection among blood donors from Texas. Ann Epidemiol. 2001 Oct;11(7):512-8. doi: 10.1016/s1047-2797(01)00242-3. PMID 11557184
- [Background] Zhang YJ, Wang XP, Deng JH, Salinas RA, Oishi N, Gao SJ. Suppression of oncogenic viral interferon regulatory factor (vIRF) of Kaposi's sarcoma-associated herpesvirus by ribozyme-mediated cleavage. Cancer Gene Ther. 2001 Apr;8(4):285-93. doi: 10.1038/sj.cgt.7700299. PMID 11393281
- [Background] Baillargeon J, Leach CT, Deng JH, Gao SJ, Jenson HB. High prevalence of human herpesvirus 8 (HHV-8) infection in south Texas children. J Med Virol. 2002 Aug;67(4):542-8. doi: 10.1002/jmv.10136. PMID 12116002
- [Background] Wang XP, Zhang YJ, Deng JH, Pan HY, Zhou FC, Gao SJ. Transcriptional regulation of Kaposi's sarcoma-associated herpesvirus-encoded oncogene viral interferon regulatory factor by a novel transcriptional silencer, Tis. J Biol Chem. 2002 Apr 5;277(14):12023-31. doi: 10.1074/jbc.M108026200. Epub 2002 Jan 30. PMID 11821384
- [Background] Zhang YJ, Pan HY, Gao SJ. Reverse transcription slippage over the mRNA secondary structure of the LIP1 gene. Biotechniques. 2001 Dec;31(6):1286, 1288, 1290, passim. doi: 10.2144/01316st02. PMID 11768657
- [Background] Wang XP, Gao SJ. Auto-activation of the transforming viral interferon regulatory factor encoded by Kaposi's sarcoma-associated herpesvirus (human herpesvirus-8). J Gen Virol. 2003 Feb;84(Pt 2):329-336. doi: 10.1099/vir.0.18653-0. PMID 12560564
- [Background] Pan HY, Zhang YJ, Wang XP, Deng JH, Zhou FC, Gao SJ. Identification of a novel cellular transcriptional repressor interacting with the latent nuclear antigen of Kaposi's sarcoma-associated herpesvirus. J Virol. 2003 Sep;77(18):9758-68. doi: 10.1128/jvi.77.18.9758-9768.2003. PMID 12941884
- [Background] Pan H, Zhou F, Gao SJ. Kaposi's sarcoma-associated herpesvirus induction of chromosome instability in primary human endothelial cells. Cancer Res. 2004 Jun 15;64(12):4064-8. doi: 10.1158/0008-5472.CAN-04-0657. PMID 15205312
- [Background] Deng JH, Zhang YJ, Wang XP, Gao SJ. Lytic replication-defective Kaposi's sarcoma-associated herpesvirus: potential role in infection and malignant transformation. J Virol. 2004 Oct;78(20):11108-20. doi: 10.1128/JVI.78.20.11108-11120.2004. PMID 15452231